CLINICAL TRIAL: NCT06556433
Title: Alaska Native Family-Based, Financial Incentives Intervention for Smoking Cessation: An RCT
Brief Title: Family-Based Financial Incentives Intervention for Smoking Cessation
Acronym: Aniqsaaq-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Alaska Native Tribal Health Consortium (Other)
Responsible Party: Principal Investigator, Christi Patten, Director, Behavioral Health Research Program, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04-015; 1R01DA056469-01A1 (NIH)
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation
Keywords: Alaska Native; Family; Financial Incentive; Smoking Cessation; Contingency Management
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rewards Group (Experimental): Index participants in the Rewards Group will be scheduled to complete smoking status check-ins six times during the 6-month Treatment Phase: weekly for four weeks, then at three and six months. At each check-in, cigarette smoking abstinence will be assessed. Participants in the Rewards Group will receive informational materials on smoking cessation.
  Interventions: Behavioral: Financial Incentive Rewards
- Comparison Group (No Intervention): Index participants in the Comparison Group will be scheduled to complete smoking status check-ins six times during the 6-month Treatment Phase: weekly for four weeks, then at three and six months. At each check-in, cigarette smoking abstinence will be assessed. Participants in the Comparison Group will receive informational materials on smoking cessation.

INTERVENTIONS:
Behavioral: Financial Incentive Rewards — Participants in the Rewards Group will have abstinence reinforced through escalating financial incentives.
  Arms: Rewards Group

SUMMARY:
The current study will conduct an RCT to evaluate the effectiveness of a family-based incentive intervention with Alaska Native/American Indian families. The experimental arm will be compared to a control arm on biochemically-confirmed smoking abstinence at 6- and 12-months post-intervention.

DETAILED DESCRIPTION:
Dyads will be stratified by the index participant's sex, and residence with family member, and by the family member's current smoking status then randomized to a no incentives control condition (n=328 dyads) or a 6-month incentive intervention (n=328 dyads).

All dyads will receive existing evidence-based cessation materials on treatment resources and social support strategies. The study will measure the index participant's smoking status in both study groups weekly during the first four weeks, and at three and six months. All participants, including support persons, will receive incentives when they complete each of the smoking status assessments. The intervention group will additionally receive individual rewards provided to the index participant for achieving verified smoking abstinence at each time point, to a maximum of $750.

The enrolled family member will also receive rewards equivalent to the value earned by the index participant that can contribute to family needs. The study will explore potential moderators (e.g., family member smoking status, index participant's sex) and mediators (e.g., interdependence) of intervention effects.

ELIGIBILITY:
Index Participant Inclusion Criteria:

* Alaska Native/American Indian (ANAI) person (based on self-reported race) and reside in Alaska.
* Age ≥18 years.
* Self-report smoking in the past 7 days, biochemically verified with saliva cotinine ≥ 30 ng/mL (positive result based on at-home saliva swab test provided by study team).
* Smoked ≥ 3 cigarettes per day over the past 3 months.
* Considering or willing to make a quit attempt.
* Have or will nominate one adult family member to enroll with them.
* Own or have access to a mobile phone or tablet with Internet and text messaging capabilities, or will be loaned an iPad for the study duration
* Willing to upload photos of self during completion of smoking status tests.
* Willing to complete and sign an Internal Revenue Service (IRS) W-9 tax identification form if they wish to receive payments on the study.
* Willing to provide written informed consent and participate in study-related tests and procedures.

Index Participant Exclusion Criteria:

* Already enrolled in the study with another family member.
* Participated in a prior study phase.

Family Member Participant Inclusion Criteria (regardless of smoking status or residence with the index participant):

* Age ≥18 years.
* Defined as family and nominated by the index participant, or have an ANAI family member who is ≥18 years and smokes that they would like to support in quitting.
* Own or have access to a mobile phone or tablet with Internet and text messaging capabilities, or will be loaned an iPad for the study duration.
* Willing to complete and sign an IRS W-9 tax identification form if they wish to receive payments on the study.
* Willing to provide written informed consent and participate in study related tests and procedures.

Both men and women, those from non-ANAI racial/ethnic groups, and those who live outside of Alaska in the United States will be eligible family member participants.

Family Member Participant Exclusion Criteria:

* Already enrolled with another family member.
* Participated in a prior study phase.

After the randomized controlled trial, qualitative interviews will be conducted with index participants, family member participants, and Alaska Tribal Health System Stakeholders to inform program implementation. Healthcare providers, cessation specialists, Elder advisors, and Tribal Health System leaders and stakeholders will be invited by the Alaska Native Tribal Health Consortium team and separately consented and interviewed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in smoking status | 6 months, 12 months
  Number of participants to have biochemically verified, prolonged smoking abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Alaska Native Tribal Health Consortium, Anchorage, Alaska, United States

REFERENCES:
- [Background] Patten CA, Koller KR, King DK, Prochaska JJ, Sinicrope PS, McDonell MG, Decker PA, Lee FR, Fosi JK, Young AM, Sabaque CV, Brown AR, Borah BJ, Thomas TK. Aniqsaaq (To Breathe): Study protocol to develop and evaluate an Alaska Native family-based financial incentive intervention for smoking cessation. Contemp Clin Trials Commun. 2023 Apr 3;33:101129. doi: 10.1016/j.conctc.2023.101129. eCollection 2023 Jun. PMID 37091507
- [Background] Sinicrope PS, Tranby BN, Young AM, Koller KR, King DK, Lee FR, Sabaque CV, Prochaska JJ, Borah BJ, Decker PA, McDonell MG, Stillwater B, Thomas TK, Patten CA. Adapting a Financial Incentives Intervention for Smoking Cessation With Alaska Native Families: Phase 1 Qualitative Research to Inform the Aniqsaaq (To Breathe) Study. Nicotine Tob Res. 2024 Sep 23;26(10):1377-1384. doi: 10.1093/ntr/ntae092. PMID 38642396
- [Background] Tranby BN, Young AM, Roche AI, Lee FR, Brown AR, Stillwater BJ, Prochaska JJ, King DK, Decker PA, Borah BJ, McDonell MG, Thomas TK, Patten CA. Beta-testing the feasibility of a family-based financial incentives smoking cessation intervention with Alaska Native families: Phase 2 of the Aniqsaaq (to breathe) Study. Contemp Clin Trials Commun. 2025 Mar 17;45:101472. doi: 10.1016/j.conctc.2025.101472. eCollection 2025 Jun. PMID 40224301